CLINICAL TRIAL: NCT05360797
Title: Randomized Multicenter Prospective Clinical Trial to Compare the Effectiveness of Home Care vs Hospital Admission in Patients With Acute Pancreatitis
Brief Title: Acute PAncreatitis and Home Care vs. Hospital Admission Study
Acronym: PADI_2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Elena Ramírez-Maldonado (Other)
Collaborators: Hospital Clinic of Barcelona (Other); Consorci Sanitari del Maresme (Other)
Responsible Party: Sponsor-Investigator, Elena Ramírez-Maldonado, Principal Investigator, Hospital Universitari Joan XXIII de Tarragona.
Organization: Hospital Universitari Joan XXIII de Tarragona. (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PADI_2
Record Dates: First submitted 2022-03-26; First posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Acute Pancreatitis; Home Care
Keywords: Pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — Hospitalization

STUDY DESIGN:
Intervention Model Description: Ramdomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Outpatient (Experimental): The Mild AP patient is discharged and contacted daily for 4 consecutive days by the study investigators in each center.
  Interventions: Other: Outpatient
- Medical home care (Experimental): The mild AP patient is discharged and contacted daily for 4 consecutive days by the medical home care department in each center.
  Interventions: Other: Medical home care
- Hospitalization (Active Comparator): The mild AP patient is hospitalized
  Interventions: Other: Hospitalization

INTERVENTIONS:
Other: Outpatient — After a 24-hour stay in the emergency department, the predictive factors of severity evaluation and the diagnosis of mild acute pancreatitis is confirmed, the patient is discharged and contacted daily for 4 consecutive days by the study investigators in each center.
  Arms: Outpatient
Other: Medical home care — After a 24-hour stay in the emergency department, the predictive factors of severity evaluation and the diagnosis of mild acute pancreatitis is confirmed, the patient is discharged and contacted daily for 4 consecutive days by the medical home care department in each center.
  Arms: Medical home care
Other: Hospitalization — After a 24-hour stay in the emergency department, the predictive factors of severity evaluation and the diagnosis of mild acute pancreatitis is confirmed, the patient is hospitalized with usual treatment (PADI_1) in each center.
  Arms: Hospitalization

SUMMARY:
Acute pancreatitis (AP) is one of the most common reason for hospitalization among gastrointestinal diseases in U.S.. The costs caused by severe AP are higher than mild AP. Nevertheless, approximately 70% of hospital admissions for AP are mild cases, if health cost saving is to be realized, it would be by lowering the cost of managing patients with mild AP without affecting patient's safety and satisfaction.

With the PADI-1 study, where it was possible to confirm the benefits of an early diet, the rapid recovery of patients with mild AP and the reduction of hospital costs, now a new scope is to be given in the treatment of patients with this pathology.

Considering the application of predictive factors of AP severity, and being sure of diagnosing mild AP, a study of home care versus hospitalization for patients with mild AP is proposed. Based on the hypothesis that outpatient care of mild AP patients would be as sage and affective as hospitalization, the aim this study is to campare the results of 3 different strategies of treatment of patients with AP mild. Additionally, satisfaction patient and costs will be analyzed.

DETAILED DESCRIPTION:
This is prospective, randomized, controlled, multicentre trial.

OBJECTIVES

Primary objective Compare the results of 3 different strategies for the management of patients with mild acute pancreatitis (AP) and to analyze differences in satisfaction patients and economic costs.

METHODS

Patients with mild AP will be randomly in three groups: group A: outpatient treatment, group B: medical home care and group C: hospitalization.

The primary and several secondary endpoints will be obtained:

1. Treatment failure rate (the primary endpoint).
2. Serum amylase, lipase, electrolytes, BUN (blood urea nitrogen), creatinine, liver function tests, and full blood count at hospital admission, 24 hours and 72 hours.
3. Relapse pain.
4. Diet intolerance.
5. Systemic complications including hemodynamic instability, renal failure, intensive care admission, surgery, radiological and endoscopic procedures.
6. Pain and Analgesic requirement.
7. Local complications including pancreatic necrosis, abscess, pseudocyst.
8. Health costs
9. Patient satisfaction

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed of AP by at least two of these three criteria: compatible abdominal pain, amylase or lipase level superior in three-fold respective laboratory baseline levels, and suitable findings in imaging techniques (CT, ultrasound or MRI).
2. age > 18 years, sign consent form.

Exclusion Criteria:

1. pregnant o breastfeeding women.
2. abdominal pain lasting >96 horas before admission.
3. the possibility of poor oral intake for reasons other than AP.
4. Pancreatic neoplasm, endoscopic retrograde cholangiopancreatography or trauma etiology, biliar obstruction.
5. Chronic pancreatitis.
6. ASA ≥3.
7. Randomization lesser the 24 hours after randomization.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
The treatment failure rate | 30 days
  Treatment failure is defined as persistence, increase or recurrence of abdominal pain, and or intolerance diet, hospital admission, and mortality

SECONDARY OUTCOMES:
Relapse of abdominal pain | 30 days
  Pain Scale: 0=No pain, 1=Very mild, 2=Discomforting, 3=Tolerable, 4=Distressing, 5=Distressing, 6=Intense pain, 7=Very intense pain, 8=Horrible pain, 9=Excruciating, 10=Unimaginable pain
Diet tolerance | 30 days
  Patient can eat at least 50% of the meals
Systemic Inflammatory Response Syndrome (SIRS) Score | 4 days
  SIRS is a simple clinical score, ranging from 0-4, that utilizes objective, routine clinical parameters (body temperature, heart rate, respiratory rate or arterial carbon dioxide tension and white blood count) that directly reflect the underlying inflammatory response. A lower change in SIRS score (negative number) indicates a better outcome (less inflammation).
Number of Participants who Development of Organ Failure | 4 days
  Including respiratory, renal and cardiovascular failures defined as modified Marshal score of equal and greater than 2. The minimum and maximum values in the modified Marshal score for each organ failure range from 0 to 4 with a higher value representing worse outcomes.
Mortality | 30 days
  Enrolled subjects that died. A death indicates a worse outcome.
Hospital admission | 30 days
  The AP patient needs hospital admission due to treatment failure
Satisfaction medical / hospital care | 30 days
  patient satisfaction is asessed comparing management with and without admittance to the hospital. Will be assessed Patient satisfaction feedback (PSF). Scale: Strongly agree, Agree, Not sure, Disagree, Strongly disagree.
Health costs | 30 days
  The costs in euros caused by diagnosis, treatment, stay in the emergency room, complications and follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Elena Ramírez-Maldonado, PhD, Principal Investigator — Hospital Universitari Joan XXIII; Rosa Jorba-Martin, PhD, Principal Investigator — Hospital Universitari Joan XXIII

IPD SHARING:
Plan to Share IPD: Yes
Study protocolo will be shared
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 01/08/2022-01/01/2023
Access Criteria: Pancreatic researchers

REFERENCES:
- [Result] Ince AT, Senturk H, Singh VK, Yildiz K, Danalioglu A, Cinar A, Uysal O, Kocaman O, Baysal B, Gurakar A. A randomized controlled trial of home monitoring versus hospitalization for mild non-alcoholic acute interstitial pancreatitis: a pilot study. Pancreatology. 2014 May-Jun;14(3):174-8. doi: 10.1016/j.pan.2014.02.007. Epub 2014 Mar 14. PMID 24854612
- [Result] Working Group IAP/APA Acute Pancreatitis Guidelines. IAP/APA evidence-based guidelines for the management of acute pancreatitis. Pancreatology. 2013 Jul-Aug;13(4 Suppl 2):e1-15. doi: 10.1016/j.pan.2013.07.063. PMID 24054878
- [Result] Greenberg JA, Hsu J, Bawazeer M, Marshall J, Friedrich JO, Nathens A, Coburn N, May GR, Pearsall E, McLeod RS. Clinical practice guideline: management of acute pancreatitis. Can J Surg. 2016 Apr;59(2):128-40. doi: 10.1503/cjs.015015. PMID 27007094
- [Result] Tenner S, Baillie J, DeWitt J, Vege SS; American College of Gastroenterology. American College of Gastroenterology guideline: management of acute pancreatitis. Am J Gastroenterol. 2013 Sep;108(9):1400-15; 1416. doi: 10.1038/ajg.2013.218. Epub 2013 Jul 30. PMID 23896955
- [Result] Yokoe M, Takada T, Mayumi T, Yoshida M, Isaji S, Wada K, Itoi T, Sata N, Gabata T, Igarashi H, Kataoka K, Hirota M, Kadoya M, Kitamura N, Kimura Y, Kiriyama S, Shirai K, Hattori T, Takeda K, Takeyama Y, Hirota M, Sekimoto M, Shikata S, Arata S, Hirata K. Japanese guidelines for the management of acute pancreatitis: Japanese Guidelines 2015. J Hepatobiliary Pancreat Sci. 2015 Jun;22(6):405-32. doi: 10.1002/jhbp.259. Epub 2015 May 13. PMID 25973947
- [Result] Ramirez-Maldonado E, Lopez Gordo S, Pueyo EM, Sanchez-Garcia A, Mayol S, Gonzalez S, Elvira J, Memba R, Fondevila C, Jorba R. Immediate Oral Refeeding in Patients With Mild and Moderate Acute Pancreatitis: A Multicenter, Randomized Controlled Trial (PADI trial). Ann Surg. 2021 Aug 1;274(2):255-263. doi: 10.1097/SLA.0000000000004596. PMID 33196485
- [Result] Pando E, Alberti P, Mata R, Gomez MJ, Vidal L, Cirera A, Dopazo C, Blanco L, Gomez C, Caralt M, Balsells J, Charco R. Early Changes in Blood Urea Nitrogen (BUN) Can Predict Mortality in Acute Pancreatitis: Comparative Study between BISAP Score, APACHE-II, and Other Laboratory Markers-A Prospective Observational Study. Can J Gastroenterol Hepatol. 2021 Mar 22;2021:6643595. doi: 10.1155/2021/6643595. eCollection 2021. PMID 33824864
- [Derived] Ramirez-Maldonado E, Rodrigo-Rodrigo M, Lopez Gordo S, Sanchez A, Coronado Llanos D, Sanchez R, Vaz J, Fondevila C, Jorba-Martin R; Catalan Pancreatitis Collaborative Group. Home care/outpatient versus hospital admission in mild acute pancreatitis: protocol of a multicentre, randomised controlled trial (PADI_2 trial). BMJ Open. 2023 Jun 28;13(6):e071265. doi: 10.1136/bmjopen-2022-071265. PMID 37380212